CLINICAL TRIAL: NCT03979547
Title: EXALT: EXercise Attenuates Liver Tumors Trial
Acronym: EXALT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jonathan Stine, Assistant Professor Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00012527
Record Dates: First submitted 2019-05-31; First posted 2019-06-07 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: perform an interventional pilot trial and randomize 21 subjects who have had a complete response to TACE to a 3-month exercise intervention (n=14) versus standard of care (n=7) where subjects are instructed to maintain their current activity level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise intervention (Experimental): The exercise program will be similar to the Exercise in All ChemoTherapy (ENACT) study which combines in-person and home-based strength training and aerobic exercise five days a week.
  Interventions: Behavioral: Exercise intervention
- Standard of Care (No Intervention): Subjects are instructed to maintain their current activity level.

INTERVENTIONS:
Behavioral: Exercise intervention — Moving Through Cancer: A Guide to Exercise for Cancer Survivors" will serve as the framework for an American College of Sports Medicine certified exercise physiologist with additional Cancer Exercise training to teach proper warm up, use of equipment, exercise form, mode of activity, intensity of exercise, flexibility exercises, and cool down.
  Arms: Exercise intervention

SUMMARY:
The overall goal of this proposal is to test the effect of exercise to delay or avert HCC recurrence and gain information regarding the potential molecular mechanisms of HCC tumor inhibition by exercise.

DETAILED DESCRIPTION:
Primary liver cancer is the leading cause of cancer worldwide. The majority of primary liver cancers are hepatocellular carcinoma (HCC) and occur in the setting of cirrhosis of the liver. Body fat and systemic inflammation are determinants of HCC risk. Cirrhotic patients with HCC are often treated with locoregional therapies including transarterial chemoembolization (TACE) as a bridge to liver transplantation. Despite this, HCC recurrence rates approach 80%. There is a growing body of evidence to suggest the benefit of exercise in cancer patients. Exercise decreases disease recurrence and improves survival in other primary cancers by altering tumor biology and influencing response to treatment. Although animal models suggest biologic plausibility, whether or not exercise prevents HCC recurrence in cancer patients remains unknown. The overall goal of this proposal is to test the effect of exercise to delay or avert HCC recurrence and gain information regarding the potential molecular mechanisms of HCC tumor inhibition by exercise.

ELIGIBILITY:
Inclusion Criteria:

* Adults age >=18 or <70 years
* Liver transplant candidates (under evaluation or listed for transplant with HCC)
* Hepatocellular Carcinoma diagnosis (HCC)
* Complete response to LRT

Exclusion Criteria:

* Active cardiac symptoms
* BMI <18 or >45 kg/m2(16)
* CPT Class B or C liver disease
* ECOG >2
* Hepatic decompensation
* Institutionalized/prisoner
* Pregnancy
* Severe medical comorbidities/psychiatric illness

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Feasibility-number of participants able to complete the trial | up to 52 weeks
  Defined as completing >80% of the sessions.(46, 47) While this would be expected for patients with cirrhosis,(46) this would be five-fold larger than the proportion of oncology patients receiving systemic treatment who complete other exercise based randomized controlled trials. We expect exercise in subjects with HCC in the background of Child Pugh Turcotte (CPT) Class A cirrhosis without hepatic decompensation (e.g., ascites, hepatic encephalopathy, bleeding gastroesophageal varices) and Eastern Cooperative Oncology Group (ECOG) 0-2 functional status to be feasible.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 52 weeks
  Data from previous oncology trials suggest up to 25% of the participants may experience a mild musculoskeletal impairment and zero adverse effects requiring treatment alterations. Pilot exercise-based trials in patients with cirrhosis have demonstrated <5% adverse events.
Acceptability-scientifically adequate | up to 52 weeks
  To assess the effectiveness of exercise trials in patients with HCC. The work with the ongoing NASHFit and completed ENACT Trials and the work of others performing exercise-based trials in patients with cirrhosis(50) has established >50% enrollment of subjects approached as a threshold of acceptability.

SECONDARY OUTCOMES:
HCC recurrence | 3- and 6- month
Overall survival | 3- and 6- month
Cancer-free survival | 3- and 6- month
waiting-list mortality | 3- and 6- month
concentration of IL-6 | 3- and 6-month
visceral adipose tissue (VAT) | 3- and 6-month
  change in body composition

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided